CLINICAL TRIAL: NCT03103282
Title: A Multi-center, Single Arm Post-market Clinical Study to Confirm Safety and Performance of PuraStat® Absorbable Haemostatic Material for the Management of Bleeding In Vascular Surgery.
Brief Title: Post-market Clinical Study to Confirm Safety and Performance of PuraStat® for the Management of Bleeding in Vascular Surgery.
Status: Completed | Type: Observational
Sponsor: 3-D Matrix Europe SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: PuraStat-002-VASC
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Vascular Anastomosis Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: PuraStat® — Synthetic haemostatic material

SUMMARY:
The objective of this post-market clinical follow-up study is to collect medical information on patients implanted with PuraStat®, according to each participating institution's procedures and standards of care.

DETAILED DESCRIPTION:
This multicentre, single arm post-market clinical study aims to collect medical information on patients implanted with PuraStat®, Absorbable Haemostatic Material, according to each participating institution's procedures and standards of care for confirming the safety and the performance of PuraStat®, for the management of bleeding in vascular surgery (Carotid Endarterectomy either by direct closure (without the use of patch), or by patch reconstruction or eversion technique).

ELIGIBILITY:
Main Inclusion criteria:

1. Male or female patient ≥18 years old
2. Subject undergoing elective carotid endarterectomy
3. Subject who is able to give voluntary, written informed consent to participate in this clinical study and from whom consent has been obtained
4. Subject, who, in the opinion of the Clinical Investigator, is able to understand this clinical study, cooperate with the study procedures and is willing to return for the required post-treatment follow-up
5. Intra-operative inclusion criteria: Subject requiring the use of PuraStat® for haemostasis during elective carotid endarterectomy either by direct closure (without the use of patch), or by patch reconstruction or eversion technique when haemostasis by ligation or standard means is insufficient or impractical.

Main exclusion criteria:

1. Presence or sequelae of coagulation disorder
2. Known allergy or hypersensitivity to any component of PuraStat®
3. Concurrent participation in another clinical trial with a medical device or a medicinal product
4. Pregnant or interested in becoming pregnant during the duration of the study, or breast feeding

   Intra-operative exclusion criteria:
5. Spurting and/or gushing haemorrhage site(s)
6. Contaminated or potentially contaminated surgical area
7. Fibrin glue and/or topical haemostatic agent used before or concomitantly to the use of PuraStat®
8. Persistent major bleeding after conventional haemostasis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective carotid endarterectomy and who have been treated with PuraStat®
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St George'S University Hospitals Nhs Foundation Trust, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- PuraStat®: Adult patients scheduled for elective carotid endarterectomy and who have been treated with PuraStat®
Period: Overall Study
Arm/Group | PuraStat®
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PuraStat®
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 53
  Belgium | 12

OUTCOME MEASURES:

1. Primary Outcome: Total Time-To-Haemostasis
Description: Total Time-To-Haemostasis (TTH) will be intraoperatively measured (secondes) from the first application of PuraStat® to a bleeding site after clamp release, until all bleeding at that site has ceased. In case of rebleeding of the treated sites and additional application of PuraStat®, the TTH will be calculated by the addition of TTH1+ TTH(n+1), where TTH1+ TTH(n+1) are the time to haemostasis after each application of PuraStat®.
Time Frame: Intraoperatively
Measure: Mean (Standard Deviation); unit: Secondes
Groups:
- PuraStat®: Adult patients scheduled for elective carotid endarterectomy and who have been treated with PuraStat® in heparin or other antiplatelet treatments during the procedure.
Arm/Group | PuraStat®
Number analyzed (Participants) | 59
Secondes | 83 (105)

2. Secondary Outcome: Status Post Application(s)
Time Frame: Intraoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | PuraStat®
Number analyzed (Participants) | 65
Participants
  Complete Haemostasis | 59
  Presence of bleeding | 6

3. Secondary Outcome: Blood Loss
Time Frame: Intraoperatively
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PuraStat®
Number analyzed (Participants) | 64
mL | 127.0 (111.4)

4. Secondary Outcome: Total Drainage Volume
Time Frame: Post-operatively
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PuraStat®
Number analyzed (Participants) | 52
mL | 50.1 (50.8)

5. Secondary Outcome: Transfusion of Blood Products
Time Frame: Intraoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | PuraStat®
Number analyzed (Participants) | 65
Participants
  NO | 63
  YES | 2

6. Secondary Outcome: Transfusion of Blood Products
Time Frame: Post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | PuraStat®
Number analyzed (Participants) | 65
Participants
  NO | 65
  YES | 0

7. Secondary Outcome: Quantity of Blood Product(s) and or Substitute(s)
Time Frame: Intraoperatively
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PuraStat®
Number analyzed (Participants) | 2
mL | 580.0 (113.1)

8. Secondary Outcome: Assessment of Product Use
Time Frame: Intraoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | PuraStat®
Number analyzed (Participants) | 65
Participants
  Ease of preparation: Excellent | 49
  Ease of preparation: Good | 16
  Ease of preparation: Fair | 0
  Ease of preparation: Poor | 0
  Ease of application: Excellent | 40
  Ease of application: Good | 25
  Ease of application: Fair | 0
  Ease of application: Poor | 0

9. Secondary Outcome: Length of Hospital Stay
Time Frame: Discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | PuraStat®
Number analyzed (Participants) | 60
Days | 4.3 (11.0)

ADVERSE EVENTS:
Time Frame: At procedure, 1 day post-operative, 5-7 days post-operative, 1 month (± 15 days) post-operative
Arm/Group | PuraStat®
All-Cause Mortality (participants affected / at risk) | 1/65
Serious Adverse Events (participants affected / at risk) | 7/65
Other Adverse Events (participants affected / at risk) | 20/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PuraStat® (N=65)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 — Events are not related to PuraStat®
Stroke (Nervous system disorders) | 3 — Events are not related to PuraStat®
Death (General disorders) | 1 — Events are not related to PuraStat®
Pneumonia (Infections and infestations) | 1 — Events are not related to PuraStat®
Bradycardia (Cardiac disorders) | 1 — Events are not related to PuraStat®
OTHER ADVERSE EVENTS (reported when occurring in more than 3.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PuraStat® (N=65)
Haemorrhage/Haematoma (Injury, poisoning and procedural complications) | 2 — AEs are related to PuraStat®
Other (Injury, poisoning and procedural complications) | 18 — AEs are not related to PuraStat®

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT03103282/SAP_000.pdf
  • Study Protocol (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT03103282/Prot_001.pdf